CLINICAL TRIAL: NCT02989714
Title: Phase Ib/II Trial of Interleukin-2 and PD-1 Checkpoint Inhibitor, Nivolumab In Metastatic Clear Cell Renal Cell Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2016.103; HUM00120502 (Other: University of Michigan)
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Interleukin-2; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HD IL2 and Nivolumab (Experimental)
  Interventions: Drug: Interleukin-2; Drug: Nivolumab

INTERVENTIONS:
Drug: Interleukin-2 — 600,000 IU/kg/dose intravenously during two 5-day cycles 9 days apart
  Other Names: High Dose Interleukin-2
Drug: Nivolumab — Nivolumab will be administered intravenously at 240 mg/dose over 60 minutes every 14 days, starting 1 week to 3 weeks after the start date of the first cycle of IL2 and continued for up to 48 weeks total in the absence of disease progression

SUMMARY:
This will be a single arm, multi-site phase Ib/II clinical trial of standard doses of High Dose Interleukin-2 (HD IL2) (600,000 IU/kg/dose intravenously during two 5-day cycles 9 days apart) in IL-2 eligible clear cell metastatic RCC (Renal Cell Carcinoma) subjects in combination with Nivolumab.

Investigators hypothesize that concurrent PD-1 inhibition synergistically enhances the anti-tumor immune response to HD IL-2 in metastatic clear cell RCC. Investigators postulate that the combination of the two therapies would result in an increase in the overall response rate, complete response rate, and improved survival outcomes compared to either of the individual therapies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histologic diagnosis of clear cell renal cell carcinoma (pure or mixed) with radiologic or histologic or cytologic evidence of metastatic disease.
* Subjects may have received up to 2 prior lines of systemic therapy (excluding any neoadjuvant/adjuvant therapy) including anti-VEGF or VEGFR inhibitor (e.g. sorafenib, pazopanib, sunitinib, bevacizumab, axitinib) or mTOR inhibitor (e.g. everolimus or temsirolimus) for metastatic disease.
* Age ≥ 18 years at the time of consent.
* ECOG (Eastern Cooperative Oncology Group) performance status (an attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 5 where 0 is asymptomatic and 5 is death.) of 0 or 1
* Adequate organ and marrow function
* Women of childbearing potential must have a negative serum or urine pregnancy test within 28 days prior to prior to registration. Women of non-childbearing potential are defined as those who have no uterus, ligation of the fallopian tubes, or permanent cessation of ovarian function due to ovarian failure or surgical removal of the ovaries. All others are considered women of child bearing potential.
* Females and males of childbearing potential must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 6 months after treatment discontinuation.
* Subjects must have measurable disease on physical exam or imaging
* An archived tissue block with the subject's renal cell carcinoma must be identified prior to registration.
* Subjects must be considered appropriate candidates for HD IL-2 by one of the treating investigators listed on the protocol. HD IL-2 candidacy evaluation is per institutional guidelines at each site and should include a dobutamine stress echocardiogram or equivalent. Subjects with a positive stress test for cardiac ischemia would be excluded from this trial.
* No clinically significant infections or any other medical condition(s) that render the subject ineligible for high dose IL-2 therapy as judged by the treating investigator.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Prior interferon or interleukin-2 therapy is NOT allowed.
* Prior anti-PD-1/PD-L1 targeted therapy is NOT allowed. Prior CTLA-4 therapy or CD40/CD40L targeted therapy is allowed.
* Prior systemic treatment must be completed at least 14 calendar days prior to registration and the subject must have recovered from the toxicities of treatment to grade 1 or better.
* Prior radiation therapy is allowed if completed at least 14 calendar days prior to registration.
* Treatment with any investigational agent or on an interventional clinical trial within 30 days prior to registration.
* No prior or concurrent malignancy is allowed except for: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, localized or locally advanced prostate cancer definitively treated without recurrence or with biochemical recurrence only, or any other cancer fully treated or from which the subject has been disease-free for at least 2 years.
* Current untreated brain metastasi(e)s. If treated history of CNS (central nervous system) metastases, should have completed radiation or surgery at least 12 weeks prior and off systemic corticosteroids.
* Autoimmune diseases such as rheumatoid arthritis are NOT allowed. Vitiligo, mild psoriasis (topical therapy only) or hypothyroidism are allowed.
* Medical need for systemic corticosteroids >10mg prednisone daily or equivalent alternative steroid (except physiologic dose for adrenal replacement therapy) or other immunosuppressive agents (such as cyclosporine or methotrexate) Topical and inhaled corticosteroids are allowed if medically needed.
* History of allergic reaction to interleukin-2 or nivolumab
* Prior history of psychiatric disorder or seizure disorders which could be exacerbated by Interleukin-2 as judged by the treating investigator. 3.2.12 Evidence of significant cardiovascular disease including history of recent (< 6 months prior) myocardial infarction, congestive heart failure, primary cardiac arrhythmias (not due to electrolyte disorder or drug toxicity, for example) beyond occasional PVC's (premature ventricular contractions), angina, positive low-level stress test, or cerebrovascular accident. All patients should have baseline pulmonary function tests. Adequate pulmonary function should be documented (FEV1 >2 liters or ≥75% of predicted for height and age) prior to initiating therapy.
* Any history of HIV or hepatitis B infection
* Any other medical or surgical condition or disease that, in the judgment of the treating physician, renders subject ineligible for High Dose Interleukin-2 therapy.
* Any history of organ allografts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2020-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajjai Alva, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (4):
- United States (4):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HD IL2 and Nivolumab
Started (Started Interleukin-2) | 13
Started Nivolumab | 12
Completed | 12
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | HD IL2 and Nivolumab
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 60 [43 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Grade 3 and Grade 4 Adverse Events of Interest
Description: This is the primary outcome for the Phase Ib portion of the trial. Events of interest are possibly immune-mediated and occur only after at least one dose of Nivolumab has been administered. Immune-mediated events of interest do not include those that are known to occur during high dose IL-2 monotherapy and are reversible. Grade assessed per CTCAE version 4.0.
Time Frame: 28 days from the first dose of Nivolumab
Population: Patients who received at least 1 dose of Nivolumab and Interleukin-2
Measure: Count of Participants; unit: Participants
Arm/Group | HD IL2 and Nivolumab
Number analyzed (Participants) | 12
Participants | 0

2. Primary Outcome: The Number of Patients That Respond to Treatment
Description: This is the primary outcome for the Phase II portion of the trial. Includes complete response (CR) + partial response (PR), measured by computerized tomography (CT) or magnetic resonance imaging (MRI) scan and assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Time Frame: 12 Weeks
Population: Patients who received at least 1 dose of Nivolumab and Interleukin-2
Measure: Count of Participants; unit: Participants
Arm/Group | HD IL2 and Nivolumab
Number analyzed (Participants) | 12
Participants | 2

3. Secondary Outcome: Number of Grade 3-5 Adverse Events of Interest
Description: Events of interest are possibly immune-mediated and occur only after at least one dose of Nivolumab has been administered. Immune-mediated events of interest do not include those that are known to occur during high dose IL-2 monotherapy and are reversible. Grade assessed per CTCAE version 4.0.
Time Frame: For the duration of the therapy plus 60 days post treatment
Population: Patients who received at least 1 dose of Nivolumab and Interleukin-2
Measure: Number; unit: events
Arm/Group | HD IL2 and Nivolumab
Number analyzed (Participants) | 12
events | 7

4. Secondary Outcome: Overall Survival at 24 Months
Description: Overall survival at 24 months following the first dose of study therapy; 24 month estimates were reported using the product limit method of Kaplan and Meier along with 95% confidence intervals.
Time Frame: 24 Months
Population: Patients who received at least 1 dose of Nivolumab and Interleukin-2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HD IL2 and Nivolumab: Interleukin-2: 600,000 IU/kg/dose intravenously during two 5-day cycles 9 days apart.
  Nivolumab will be administered intravenously at 240 mg/dose over 60 minutes every 14 days, starting 1 week to 3 weeks after the start date of the first cycle of IL2 and continued for up to 48 weeks total in the absence of disease progression.
Arm/Group | HD IL2 and Nivolumab
Number analyzed (Participants) | 12
percentage of participants | 77.1 [34.5 to 93.9]

5. Secondary Outcome: Progression Free Survival (PFS) at 24 Months
Description: PFS is defined as the time from start of study therapy with Nivolumab until progression or death; up to 24 months. Progressive disease is defined as At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions.
Time Frame: 24 Months
Population: Patients who received at least 1 dose of Nivolumab and Interleukin-2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HD IL2 and Nivolumab
Number analyzed (Participants) | 12
percentage of participants | 43.6 [14.7 to 69.9]

ADVERSE EVENTS:
Time Frame: 60 days after end of treatment (Up to 14 months)
Arm/Group | HD IL2 and Nivolumab
All-Cause Mortality (participants affected / at risk) | 2/13
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HD IL2 and Nivolumab (N=13)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HD IL2 and Nivolumab (N=13)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 11 (36)
Alkaline phosphatase increased (Investigations) | 8 (16)
Allergic reaction (Immune system disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 11 (25)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 11 (33)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 9 (18)
Cardiac troponin T increased (Investigations) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 10 (18)
Chronic kidney disease (Renal and urinary disorders) | 1 (4)
Colitis (Gastrointestinal disorders) | 2 (2)
Confusion (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
CPK increased (Investigations) | 1 (3)
Creatinine increased (Investigations) | 9 (35)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (18)
Dizziness (Nervous system disorders) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Dysphasia (Nervous system disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 6 (6)
Encephalopathy (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Eye disorders - Other (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Fatigue (General disorders) | 11 (14)
Fever (General disorders) | 3 (4)
Flushing (Vascular disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (42)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (11)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (35)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (34)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 4 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 7 (12)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Hypotension (Vascular disorders) | 10 (16)
Hypothyroidism (Endocrine disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 8 (32)
Lymphocyte count increased (Investigations) | 5 (10)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (16)
Neutrophil count decreased (Investigations) | 2 (3)
Oral pain (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Papulopustular rash (Infections and infestations) | 4 (4)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 8 (20)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (20)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 4 (5)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Urine output decreased (Investigations) | 3 (5)
Vaginal infection (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (14)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 4 (10)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial did not meet criteria for continuation to the second stage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT02989714/Prot_SAP_000.pdf